## Janssen Research & Development \*

## Addendum to the Statistical Analysis Plan

A Phase 3 Randomized, Placebo-controlled Double-blind Study of JNJ-56021927 in Combination with Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Subjects with Metastatic Castration-resistant Prostate Cancer (mCRPC)

#### Protocol 56021927PCR3001; Phase 3

#### JNJ-56021927

\*Janssen Research & Development is a global organization that operates through different legal entities in various countries. Therefore, the legal entity acting as the sponsor for Janssen Research & Development studies may vary, such as, but not limited to Aragon Pharmaceuticals Inc, Janssen Biotech, Inc.; Janssen Products, LP; Janssen Biologics, BV; Janssen-Cilag International NV; Janssen, Inc; Janssen Infectious Diseases BVBA; Janssen R&D Ireland; or Janssen Research & Development, LLC. The term "sponsor" is used throughout the protocol to represent these various legal entities; the sponsor is identified on the Contact Information page that accompanies the protocol.

**Status:** Approved

Date: 21 September 2020

**Prepared by:** Janssen Research & Development, LLC

**Document No.:** EDMS-RIM-146748, 1.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

## **BACKGROUND AND RATIONALE**

At the first and second interim analysis of the study (for overall survival), the IDMC has recommended that the study continue without modification, continue to collect data on all the secondary endpoints and remain blinded until the final analysis of OS. This addendum provides clarification on the data sources in this study that will be used in the primary analysis (and the relevant sensitivity analyses) for the secondary endpoint of CCI



## SECONDARY ENDPOINT OF TIME TO PAIN PROGRESSION

The main feature of this addendum to the SAP for the final analysis is to include the CRF in addition to that described in the original SAP which included patient reported BPI3 worst pain score and the use of chronic opioid, whichever occurs first.

An additional sensitivity analysis of this endpoint is included in this addendum that incorporates selected deaths as pain progression events. Specifically, a death event meeting at least one of the CCI

#### FINAL ANALYSIS OF SECONDARY ENDPOINTS IN GROUP 1



## **BIOMARKER SUBGROUP ANALYSIS**

Additional biomarker analyses are also pre-specified in this addendum based on the most recent tumor analysis findings from the two unblinded apalutamide phase 3 trials, SPARTAN and TITAN, using CCI.



each treatment arm. Association with time to event endpoints will be evaluated using

## Janssen Research & Development \*

## **Statistical Analysis Plan**

A Phase 3 Randomized, Placebo-controlled Double-blind Study of JNJ-56021927 in Combination with Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Subjects with Metastatic Castration-resistant Prostate Cancer (mCRPC)

### Protocol 56021927PCR3001; Phase 3

#### JNJ-56021927

\*Janssen Research & Development is a global organization that operates through different legal entities in various countries. Therefore, the legal entity acting as the sponsor for Janssen Research & Development studies may vary, such as, but not limited to Aragon Pharmaceuticals Inc, Janssen Biotech, Inc.; Janssen Products, LP; Janssen Biologics, BV; Janssen-Cilag International NV; Janssen, Inc; Janssen Infectious Diseases BVBA; Janssen R&D Ireland; or Janssen Research & Development, LLC. The term "sponsor" is used throughout the protocol to represent these various legal entities; the sponsor is identified on the Contact Information page that accompanies the protocol.

Status: Approved

**Date:** 31 October 2018

**Prepared by:** Janssen Research & Development, LLC

**Document No.:** EDMS-ERI-162095981, 2.0

**Compliance:** The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable law or regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you that is indicated as privileged or confidential.

# **TABLE OF CONTENTS**

| TAB | BLE OF CONTENTS | <u>2</u> |
|-------|---------------------------------------------------------|----------|
| AMI | ENDMENT HISTORY | 4 |
| ABB | BREVIATIONS | 5 |
| 1. | INTRODUCTION | 7 |
| 1.1. | Trial Objectives | 7 |
| 1.1.1 | 1. Primary Objective | 7 |
| 1.1.2 | 2. Secondary Objectives | 7 |
| 1.1.3 | 3. Other Objectives | 7 |
| 1.2. | Trial Design | 7 |
| 1.3. | Statistical Hypotheses for Trial Objectives. | 8 |
| 1.4. | r | |
| 1.5. | | |
| 1.5.1 | | |
| 1.5.2 | 2. Blinding | 9 |
| 2. | GENERAL ANALYSIS DEFINITIONS | 0 |
| 2.1. | | |
| 2.2. | · · · · · · · | |
| 2.3. | 5 | |
| 2.4. | J = | |
| 2 | INTERIM ANALYSIS AND INDEPENDENT DATA MONITORING COMMIT | |
| 3. | REVIEW | |
| 3.1. | | |
| 3.1.1 | <b>,</b> | |
| 3.1.2 | | |
| 3.2. | <b>,</b> | |
| 4. | SUBJECT INFORMATION | 12 |
| 4.1. | | |
| 4.2. | | |
| 4.3. | * | |
| 4.4. | <u>.</u> | |
| 4.5. | Prior and Concomitant Medications | |
| 4.6. | Subsequent Anti-cancer Therapies | 14 |
| 5. | EFFICACY | 14 |
| 5.1. | | |
| 5.1.1 | $\mathcal{I}$ | |
| 5.1.2 | | |
| 5.2. | Primary Endpoint of rPFS. | |
| 5.2.1 | | |
| 5.2.2 | | |
| 5.2.3 | <b>,</b> | |
| 5.2.4 | | |
| 5.3. | | |
| 5.3.1 | • • | |
| 5.3.2 | | |

| 5.3.3.<br>5.4.<br>5.4.1.<br>5.4.2.<br>5.4.3. | Other Efficacy Analyses Definition Analysis Methods | 21<br>21<br>23 |
|---|---|---|
| 6. | SAFETY | 23 |
| 6.1. | Adverse Events | |
| 6.2. | Clinical Laboratory Tests | 25 |
| 6.3. | Vital Signs and Physical Examination Findings | |
| 6.4. | Electrocardiogram | 26 |
| 7. | PHARMACOKINETICS | 26 |
| 8. | BIOMARKERS | 26 |
| 9. | MEDICAL RESOUURCE UTILIZATION | 27 |
| REF | ERENCES | 28 |
| | chment 1: Audit Analysis Using Amit's Method | |
| Attac | chment 2: Adverse Events of Special Interest or Clinical importance | 31 |
| TAB | ILES | |
| Table | e 1: Key censoring Rule | 16 |
| Table | | |
| Table | e 3: Other Endpoints | |
| Table | $\iota$ | |
| | Progression | 29 |

# AMENDMENT HISTORY

| SAP Version | Issue Date |
|-------------|-------------|
| Original | 3 May 2018 |
| Amendment 1 | 31 Oct 2018 |

# Amendment 1 (31 October 2018)

The rationale for and description of the changes are listed below, when revisions are provided verbatim, bold font denotes new text, and strikethrough denotes deleted text.

| Applicable Section(s) | Description of Change(s) |
|---|---|
| Section 5.3.1 | Rationale: |
| Secondary endpoints definition | The secondary endpoints (time to pain progression and time to chronic opioid use) are assessed from time of randomization to pain progression (as defined in Section 5.3.1) and to time to chronic opioid use (as defined in Section 5.3.1). The original text regarding censoring in the last paragraph of Section 5.3.1 has been amended to clarify that censoring for subsequent therapy was intended as an additional sensitivity analysis for these endpoints. Original text: Additionally, for time to chronic opioid use and time to pain progression endpoints, the initiation of anti-cancer subsequent therapy will be used to censor the event after the therapy. Replaced with: Additionally, sensitivity analyses will be performed for time to chronic opioid use and time to pain progression endpoints, the initiation of anti-cancer subsequent therapy will be used to censor the event after the therapy. |

#### **ABBREVIATIONS**

AA abiraterone acetate

AAP abiraterone acetate plus prednisone or prednisolone

ADT androgen deprivation therapy

AE adverse event ALB albumin

ALK-P alkaline phosphatase
ALT/SGPT alanine aminotransferase
ANC absolute neutrophil count
ANCOVA analysis of covariance
AR androgen receptor

AST/SGOT aspartate aminotransferase

BICR Blinded Independent Central Review

BID twice daily

BPI-SF Brief Pain Inventory-Short Form

CI confidence interval CRF case report form

CRO Contract Research Organization
CRPC castration-resistant prostate cancer

CSR Clinical Study Report CT computed tomography

CTCAE Common Terminology Criteria for Adverse Events

DHEA-S dihydroepiandrosterone sulphate DMC Data Monitoring Committee

ECG Electrocardiogram

ECOG Eastern Cooperative Oncology Group

eCRF electronic case report form

EU European Union

FACT-P Functional Assessment of Cancer Therapy – Prostate

FDA Food and Drug Administration GnRH gonadotropin releasing hormone

HDL high density lipoprotein

HR hazard ratio

ICH International Conference on Harmonization IDMC Independent Data Monitoring Committee

ITT Intent-to-Treat

LE Investigator or local site evaluation (imaging)

IWRS Interactive Web Response System LOCF last observation carried forward

LDH lactate dehydrogenase LDL low density lipoprotein

LHRH luteinizing hormone-releasing hormone
MedDRA Medical Dictionary for Regulatory Activities

MRI magnetic resonance imaging MRU medical resource utilization NCI National Cancer Institute

OS overall survival

PCWG2 Prostate Cancer Working Group

PD Phgroupacodynamic
PI principal investigator
PK phgroupacokinetic(s)
PRO patient-reported outcome
PS performance status
PSA prostate specific antigen

PT preferred term QD once daily

| RECIST | Response | Evaluation | Criteria | in Solid | Tumors |
|--------|----------|------------|----------|----------|--------|

ROW Rest of World

rPFS radiographic progression-free survival

SAE serious adverse event
SAP Statistical Analysis Plan
SD standard deviation
SOC system organ class

SSRE symptomatic skeletal-related event

TLGs tables, listings, and graphs ULN upper limit of normal

US United States

WHO World Health Organization

#### 1. INTRODUCTION

This document describes the planned statistical analyses for Protocol 56021927PCR3001: A Phase 3 Randomized, Placebo-controlled Double-blind Study of JNJ-56021927 in Combination with Abiraterone Acetate and Prednisone Versus Abiraterone Acetate and Prednisone in Subjects with Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer (mCRPC). This statistical analysis plan (SAP) is intended to supplement the study protocol. Any deviations from this analysis plan will be described in the clinical study report.

## 1.1. Trial Objectives

## 1.1.1. Primary Objective

The primary objective is to compare the radiographic progression-free survival (rPFS) of apalutamide in combination with abiraterone acetate (AA) plus prednisone or prednisolone (AAP) and AAP in subjects with chemotherapy-naïve mCRPC.

## 1.1.2. Secondary Objectives

The secondary objectives of this study are:

- To characterize the safety profile of apalutamide in combination with AAP
- To characterize the population pharmacokinetics (PK) of apalutamide and abiraterone

## 1.1.3. Other Objectives

The other objectives of this study are:

- To explore the relationship between PK and pharmacodynamics (PD) of apalutamide and abiraterone
- To evaluate exploratory biomarkers predictive of response and resistance in subjects when treated with apalutamide in combination with AAP compared with AAP
- To assess the effect on patient-reported outcomes (PROs) in this study population when treated with apalutamide in combination with AAP compared with AAP
- To evaluate other endpoints of clinical relevance including additional assessments of pain, objective response, time to symptomatic skeletal-related event (SSRE), and PSA response
- To evaluate medical resource utilization information (MRU)

## 1.2. Trial Design

This is a randomized, double-blind placebo-controlled, multinational, multicenter Phase 3 study to determine if subjects with chemotherapy-naïve mCRPC will benefit from the addition of apalutamide to AAP compared with AAP. Subjects will continue ADT (in this study, GnRHa or surgical castration). Approximately 960 subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive apalutamide and AAP or matching placebo and AAP. Subjects will be stratified by the presence or absence of visceral metastases, Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) grade of 0 or 1, and region (European Union [EU], North America [United States/Canada], and Rest of World [ROW]). The study will consist of a Screening Phase; a

Treatment Phase, and a Followup Phase. The study is anticipated to end approximately 84 months after the first subject is randomized. A study design scheme is provided in protocol Figure 2.

A treatment cycle is defined as 28 days. Treatment will continue until disease progression, unacceptable toxicity, death or the sponsor terminates the study. Subjects must discontinue study drugs with documented unequivocal clinical progression (protocol Section 10.2). If the subject has radiographic progression, but not unequivocal clinical progression, and alternate treatment is not initiated, the subject may continue on study treatment at the investigator's discretion.

After discontinuing study drug, subjects will be contacted every 3 months (protocol Section 9.1.5) until death or termination of the study. In addition to survival follow up, analgesic use, SSREs, ECOG PS, and subsequent therapy for prostate cancer up to and including chemotherapy will be collected. Patient-reported outcomes (PROs) questionnaires will also be administered every 3 months for up to 12 months after treatment discontinuation.

Subjects will be monitored for safety during the Screening and Treatment Phases and up to 30 days after the last dose of study drug. Adverse events, including clinically significant laboratory abnormalities reported as AEs, will be graded and summarized using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.03. Dose modification guidelines will be provided.

## 1.3. Statistical Hypotheses for Trial Objectives

The primary hypothesis of the study is that apalutamide in combination with AAP compared with AAP will demonstrate improved rPFS and an acceptable safety profile in subjects with chemotherapy-naïve mCRPC. The statistical hypothesis is listed as follows:

 $H_0$ : The rPFS distributions of the combination group (apalutamide+AAP),  $S_A(t)$ , and that of the control group (Placebo+AAP),  $S_P(t)$ , are equal:

$$S_A(t) = S_P(t)$$
, for all  $t > 0$ 

H<sub>1</sub>: The rPFS distributions are not equal for at least one time point t:

$$S_A(t) \neq S_P(t)$$
, for some  $t > 0$ 

where rPFS is defined as the time from the date of randomization to the date of radiographic progression or death, whichever occurs first. Radiographic progression for primary endpoint will be based on the investigator's assessment of soft tissue lesion using computed tomography (CT)/magnetic resonance imaging (MRI) per response evaluation criteria in solid tumors (RECIST 1.1)<sup>[1]</sup> and bone lesion progression on bone scans per modified Prostate Cancer Working Group 2 (PCWG2)<sup>[2]</sup>.

## 1.4. Sample Size Justification

This study is designed to provide sufficient power (approximately of the control group in the secondary endpoint of OS based on an assumed median OS of of the control group (AAP). The assumption for OS is a HR of the control group of the control group of apalutamide plus AAP compared with the control group of AAP alone. Under the assumption that the failure distribution of OS follows an exponential distribution with a constant HR, approximately death events will be required to detect the assumed HR at a maximum two-sided significance level of

0.05, with enrollment duration of approximately (approximately 960 subjects) and additional follow-up of CCI to reach the total number of events. The median time of OS in the control group of AAP alone and the enrollment projection are assumed based on the observation in the COU-AA-302 study. See Section 5.3 for detail statistical procedure use in the adjustment of the significance level for OS.

It is assumed that the failure distribution of the primary endpoint, rPFS follows an exponential distribution with a constant hazard rate. The assumption for rPFS is a hazard ratio of color, a % risk reduction of experiencing radiographic progression or death. This represents an improvement in the median time to radiographic progression or death of approximately colored longer in the treatment group of apalutamide plus AAP than in the control group of AAP alone. Based on simulation to account for the correlation between rPFS and OS, it is estimated that approximately rPFS events would be required to provide at least power in detecting a hazard ratio (HR) of colored (median rPFS) of for the control group [AAP] versus for the treatment group [apalutamide and AAP] at a two-sided significance level of 0.05 under the assumption of a positive correlation between rPFS and OS (r = colored (rPFS)). The median time of rPFS in the control group of AAP alone and the correlation between rPFS and OS are assumed based on the observation in the COU-AA-302 study. The same enrollment assumptions as described for OS are assumed.

### 1.5. Randomization and Blinding

#### 1.5.1. Randomization

Subjects who meet all the inclusion criteria and none of the exclusion criteria will be randomized in a 1:1 ratio to receive apalutamide and AAP or matching placebo and AAP using permuted block randomization. Subjects will be stratified by:

- Visceral metastases (Presence vs. absence)
- ECOG performance status (Grade of 0 or 1)
- Region (EU, NA, and ROW)

The countries included in each region are listed as below. NA: US and Canada; EU: Belgium, France, Germany, Italy, Netherlands, Spain, and UK; ROW: Australia, Korea, China, Japan, South Africa, Russia, Mexico, Brazil, and Argentina.

## 1.5.2. Blinding

This study is a double blind study. All subjects and study team members associated with the study conduct are to remain blinded to treatment group assignment until the time of database lock and unblinding of the study. Unblinding during the study can only happen in the case of a safety or a medical emergency, or for conducting data review by the IDMC as outlined in the IDMC charter.

#### 2. GENERAL ANALYSIS DEFINITIONS

**Study Day**: For safety, study day will be calculated in reference to the date of first dose. Study Day 1 corresponds to the date the subject receives first dose of study drug. For Efficacy analysis, Study day will be calculated in reference to the date of randomization.

**Cycle**: For the purpose of the study, a treatment cycle is defined as 28 days. Subjects will begin taking study drug on Day 1 of Cycle 1.

**Baseline Value**: Unless otherwise specified, the baseline value will be defined as the closest measurement prior to the first dose of study drug. Change from baseline will be defined as (post-baseline value – baseline value).

**Treatment Duration**: Treatment duration will be defined as the duration of time from the date of the first dose of study drug to the date of last dose of study drug.

**Time to event**: Time to event calculations will be defined as the time from randomization to the date of the event of interest. Time to event or duration of event endpoints will be based on the actual date of the event, not visit number or visit label.

#### 2.1. Visit Windows

The Treatment Phase will begin at Cycle 1 Day 1 of treatment and will continue until study drug is discontinued. Subjects should start study drug within 72 hours after randomization. Visits for each cycle will have a  $\pm 2$  day window.

Subjects' time on study will be determined in Study Days. Study Day 1 will be defined as the first day of dosing. Positive study days will count forward from Study Day 1. Study Day -1 will be the day before Study Day 1, and all subsequent negative study days will be measured backward from Study Day -1. There will be no Study Day 0. The last available value collected prior to the first dose of study drug will be used as the baseline value.

Study Day will be used in the analysis of safety data. The protocol allows a 72-hour window (3 calendar days) between randomization and the first dose; all efficacy analyses on time-to-event endpoints will consider the date of randomization as Day 1.

#### 2.2. Pooling Algorithm for Analysis Centers

There is no plan for pooling the centers (study sites) for efficacy or safety analyses, unless analysis by site is warranted.

## 2.3. Analysis Sets

The following analysis sets will be used for this study:

Intent-to-Treat (ITT) Population: The ITT population includes all randomized subjects and will be classified according to their assigned treatment group, regardless of the actual treatment received. Subject disposition and efficacy analyses will be performed on data from the ITT population.

Safety Population: The safety population includes all subjects who received at least 1 dose of study drug as actually treated.

Patient-report Outcomes Population [PRO]: The PRO population includes all randomized subjects who completed at least the baseline assessment of the BPI-SF, FACT-P or EQ-5D-5L questionnaires. All time-to-event analysis will be based on ITT population.

Population Pharmacokinetics Populations [PK]: The PK population includes all randomized subjects who have at least 1 PK sample collected.

Biomarker Population: All randomized subjects who have at least 1 biomarker sample collected.

## 2.4. Definition of Subgroups

In order to assess the consistency of treatment benefit with respect to the primary efficacy endpoint of rPFS and the secondary endpoint of OS, additional univariate analyses will be performed for the following important subgroups:

- Baseline ECOG performance status (0, 1)
- Presence of visceral metastases (yes, no)
- Baseline Brief Pain Inventory-Short Form (BPI-SF) Question 3 (worst pain in the last 24 hours) score (0 to  $\le 1, >1$  to  $\le 3, >3$ )
- Bone metastasis only at entry (yes, no)
- Number of bone lesions at baseline (<=10 vs. >10)
- Age  $(<65, \ge 65, \ge 75)$
- Baseline PSA above median (yes, no)
- Baseline LDH above median (yes, no)
- Baseline ALP above median (yes, no)
- Geographic region (EU, NA, ROW)

Subgroup analysis of selected countries will be performed for regional regulatory filing purpose.

# 3. INTERIM ANALYSIS AND INDEPENDENT DATA MONITORING COMMITTEE REVIEW

#### 3.1. Interim Analysis

#### 3.1.1. Futility Analysis

A non-binding futility analysis using an intermediate endpoint, the prostate-specific antigen (PSA) 90% decline rate (PSA90), is planned when approximately subjects have been treated for at least cycles. The PSA90 is defined as  $\geq$  90% maximum decrease in PSA from baseline. Under the assumption of a correlation between PSA90 and OS of observed in the COU-AA-302 study, a clinically meaningful improvement from decline rate in the control group to subjects will be required. The study may be considered futile if the p-value obtained from a chi-square test is color. The purpose of this analysis is to provide an early look at PSA90 to ensure that the combination of apalutamide plus AAP has sufficient antitumor activity compared with AAP. This futility analysis will not be used to substantiate an efficacy claim.

A non-binding futility analysis using rPFS will be implemented after observing color (color events) of the total number of required color events. The study may be considered futile if the estimated hazard ratio (HR) from Cox proportional-hazard model is greater than color than the probability of stopping under null hypothesis is color and the probability of stopping under alternative hypothesis is color.

Non-binding futility analyses are also being implemented for the OS endpoint (see Section 5.3, Table 2).

## 3.1.2. Interim Analysis

There will be no interim analysis of the primary rPFS endpoint.



## 3.2. Independent Data Monitoring Committee (IDMC)

An IDMC will be commissioned for the study to perform regular safety review and the planned interim analyses. The IDMC will review the safety data when the first 60 subjects who have completed at least 1 cycle of treatment.

The IDMC will review the progress of the study and cumulative masked (ie, A vs B instead of actual treatment designation) safety data on a periodic basis as well as serve as the primary reviewer of the efficacy analyses.

Complete details regarding the composition and governance of the IDMC will be outlined in the IDMC Charter.

#### 4. SUBJECT INFORMATION

## 4.1. Demographics and Baseline Characteristics

The following parameters will be summarized by treatment group and overall using the ITT population:

- Age, sex, race, ethnicity, weight, height
- Baseline ECOG performance status
- Baseline PSA value
- Baseline Hemoglobin value
- Baseline Lactate Dehydrogenase value
- Baseline Alkaline Phosphatase value
- Baseline Testosterone value
- Average of 7-day BPI-SF Pain Score (Q3) leading to Cycle 1 Day 1 (with minimum 1 day)
- Baseline Analgesic Usage Score
- Time from Initial Diagnosis to First Dose
- Tumor Stage at Diagnosis
- Lymph Node Stage at Diagnosis
- Gleason Score at Initial Diagnosis

#### Extent of Disease

## 4.2. Disposition Information

Subject enrollment and disposition will be summarized by treatment group. The summary of subject disposition will display the number of subjects screened, the number of subjects who screen failed, the number of subjects randomized, and the number of subjects in the ITT, safety, and population PK populations. The summary will also include the number and percent of subjects who are ongoing in the treatment and who discontinued from treatment and reason for discontinuation.

## 4.3. Treatment Compliance and Extent of Exposure

The safety population will be used to summarize drug exposure, treatment compliance, and dose modifications by treatment group.

Treatment duration will be defined as the duration from the date of the first dose of study drug to the date of last dose of study drug. The number of tablets taken will be calculated based on the number of tablets dispensed at the study visits minus the number of returned tablets.

The percent overall treatment compliance will be defined as the number of tablets taken during the study divided by the expected number of tablets, multiplied by 100. Each subject should be taking a maximum of 8 tablets of study drug (excluding prednisone) per day while on the study. A subject's expected number of tablets will be calculated as the number of assigned tablets per day multiplied by treatment duration.

Subjects with at least one dose modification and the reason for the dose modification will be summarized by treatment group.

#### 4.4. Protocol Deviations

Protocol deviations and eligibility deviations will also be summarized by treatment group. Protocol deviations will be reviewed on a case-by-case basis and assessed if they are considered major deviations for this study. The final list will be complied prior to database lock. The major protocol deviations may include, but are not limited to, the following:

- Deviation from inclusion/exclusion criteria that may affect efficacy endpoints
- Major study drug dosing errors or dose modifications that are not within the protocol specifications that may compromise subject safety or efficacy assessments.
- Administration of prohibited concomitant medication during the course of the study treatment period
- Any other deviation that impacts subject safety

#### 4.5. Prior and Concomitant Medications

Prior and concomitant medications, other than study treatment, taken prior to starting study treatment and those administered during the study will be summarized by treatment group. Medications are considered concomitant if taken during the treatment period (within 30 days of the last study drug dose). Medications will be summarized by WHO Drug therapeutic class and generic medication name.

## 4.6. Subsequent Anti-cancer Therapies

Subsequent therapies received after discontinuation of study treatment will be summarized by treatment arm in the overall population as well as by geographic region.

The following imputation rule will be used for missing start dates for subsequent therapies:

- a. If all parts of the start date are missing, the date will be imputed with the date after the discontinuation date.
- b. In the case where only the start day of therapy is missing, it will be replaced by the day after the discontinuation date if the therapy starts in the same month and year as the discontinuation date. Otherwise, it will be replaced by the first of the month.

If both the start day and month of therapy are missing, the start day and month will be replaced by the day and month of the date after the discontinuation date if the therapy and the discontinuation occur in the same year; otherwise, it will be replaced by 1<sup>st</sup> of January.

#### 5. EFFICACY

This section outlines the planned analyses of the primary and secondary efficacy, and other endpoints of the study

Efficacy analyses will be performed in the ITT population, incorporating the randomization stratification factors as documented on the electronic case report form (eCRF) from the interactive web response system (IWRS), unless otherwise specified. All continuous variables will be summarized using number of subjects (n), mean, standard deviation (SD), median, minimum, and maximum. Categorical variables will be summarized with count and percentage.

Time-to-event endpoints will be summarized using the Kaplan-Meier method<sup>[5]</sup> and displayed graphically where appropriate. Median event times and two-sided 95% confidence interval (CI) for each treatment group will be provided. Stratified Cox proportional-hazard models will be used to estimate the HR and its 95% CI. The stratification factors to be used in the model are presence or absence of visceral metastases, ECOG performance status, and region.

The testing for the time-to-event endpoints will be based on the stratified log rank test; non-stratified log rank test will be performed as a sensitivity analysis, as appropriate. Multivariate Cox regression analysis, adjusting for important selected prognostic factors, will be performed as supportive analyses for rPFS and OS. The details of including prognostic factors can be found in Section 5.2.4 and additional exploratory analysis can be found in Section 5.3.3.

The proportional hazard assumption will be assessed graphically by plotting log (-log [estimated survival distribution function]) against log (survival time). The resulting graphs should have approximately parallel lines when the assumption holds. If the proportional hazards assumption is reasonably met, then the HR will be used as an estimate of treatment effect. If the proportional hazards assumption is violated, then the inference remains statistically valid for testing equality in survival distributions, but treatment effect will only be estimated using the median time to event in each treatment group.

Endpoints with binary outcome (e.g., objective response rate) will be summarized by descriptive statistics (count and percentage) by the treatment group. The relative risk (treatment: control) will be reported along with the corresponding two-sided 95% CI. The response rates between two treatment groups will be

compared by using the chi-square test; Fisher's exact test may be used if the expected counts in some of the cells are less than 5.

## 5.1. Analysis Specifications

## **5.1.1.** Level of Significance

In general, a two-sided significance level of  $\alpha = 0.05$  will be used for all hypothesis testing and all confidence intervals will be calculated on the two-sided 95% confidence level, unless otherwise specified.

# **5.1.2.** Data Handling Rules

In general, no imputation method is planned for handling missing or incomplete data unless specified otherwise for a specific endpoint. Sensitivity analyses with censoring rules may be conducted if warranted and will be documented in the clinical study report.

The following imputation rule will be used for missing dates in the assessment of an event:

- a. If all parts of the date are missing, the date will not be imputed.
- b. In the case where only the start day of an event is missing, it will be replaced by the start day of study treatment if the event occurs in the same month and year. Otherwise, it will be replaced by the first date of the month.
- c. If the stop day is missing, the stop day of the event will be replaced by the stop day of study treatment. Otherwise, the last day of the month will be used to replace the missing stop day.
- d. If both the start day and month of an event are missing, the start day and month will be replaced by the start day and month of study treatment if the event and the start of the treatment occur in the same year; otherwise, it will be replaced by 1<sup>st</sup> of January.

If both the stop day and month of an event are missing, the stop day and month will be replaced by the stop day and month of study treatment if the event and the stop of the treatment occur in the same year; otherwise, it will be replaced by 31<sup>st</sup> of December.

## 5.2. Primary Endpoint of rPFS

#### 5.2.1. Definition

The primary efficacy endpoint is radiographic progression-free survival (rPFS), based on the imaging assessments by the investigator, is defined as the time from the date of randomization to the date of first documentation of radiographic progressive disease or death due to any cause, whichever occurs first.

Radiographic progression in this study is defined as the time from randomization to the occurrence of one of the following:

- A subject is considered to have progressed by bone scan if:
  - The first bone scan with  $\ge 2$  new lesions compared with baseline is observed <12 weeks from randomization and is confirmed by a second bone scan taken  $\ge 6$  weeks later showing  $\ge 2$  additional new lesions (a total of  $\ge 4$  new lesions compared with baseline);

- The first bone scan with  $\ge 2$  new lesions compared with baseline is observed  $\ge 12$  weeks from randomization and the  $\ge 2$  new lesions are verified on the next bone scan  $\ge 6$  weeks later (a total of  $\ge 2$  new lesions compared with baseline).
- Progression of soft tissue lesions measured by computed tomography (CT) or magnetic resonance imaging (MRI) as defined in modified RECIST 1.1 criteria.

Subjects that withdraw from the study (i.e., withdrawal of consent, lost to follow-up) or receive new systemic anti-cancer therapy without documented disease progression will be censored on the date of the last tumor assessment. Subjects with no evidence of radiographic progressive disease or death will be censored on the date of the last tumor assessment. If there was no tumor assessment performed after the baseline visit, the subject will be censored on the date of randomization. Key censoring rules are summarized as shown in Table 1. More detailed censoring rules are documented in Data Presentation Specifications (DPS).

**Table 1:** Key censoring Rule

| Scenario | Censoring rule |
|---|---|
| No tumor assessment at Baseline | Censored on the date of randomization |
| or | |
| No tumor assessment after Baseline | |
| Subjects who are lost to follow-up or withdraw from study | Censored on the date of the last tumor |
| | assessment |
| Subjects who receive new systemic anti-cancer therapy prior to | Censored on the date of the last tumor |
| documented disease progression or death | assessment prior to the start of the new |
| | systemic anti-cancer therapy |
| Subjects with no evidence of radiographic progressive disease | Censored on the date of the last tumor |
| or death | assessment |
| Subjects who miss ≥2 consecutive planned radiographic scans | Censored on the date of the last tumor |
| or has ≥2 consecutive unreadable scans before progression or | assessment before the |
| death | missed/unreadable scans |

## 5.2.2. Analysis Methods

The primary analysis for the comparison of the survival distributions of rPFS between two treatment groups will be carried out using the stratified log rank test at a two-sided significance level of 0.05. If the number of events required for the primary analysis of rPFS and the first interim analysis of OS occur approximately at the same time, the primary analysis of rPFS will be performed at the time of the first interim analysis of OS. Otherwise, the timing of the primary analysis of rPFS may be adjusted taking into consideration the number of death events.

Non-stratified log rank test will be performed as a sensitivity analysis. Stratified Cox proportional-hazard model will be used to obtain the HR and its 95% confidence interval.

#### 5.2.3. Audit Plan

In this study, the primary efficacy endpoint of rPFS is based on the investigators' radiographic evaluation of the disease. To confirm that the investigator or local site evaluation (LE) is not biased in favor of the experimental arm, an audit plan based on the NCI method (Dodd et.al., Biometrics) <sup>[6]</sup> will be implemented. This plan includes a subset of subjects randomly selected for a blinded independent central review (BICR).

The goal of the audit method by Dodd et al is to provide confidence that the local site evaluation of any treatment effect for rPFS is a true estimate and unlikely to be affected by investigator bias. Assuming an observed investigator-assessed HR for rPFS of 0.5-0.75, an audit size of approximately 60% of all randomized subjects is recommended by Dodd et.al. (Biometrics 2011)<sup>[6]</sup> and Zhang (2013)<sup>[8]</sup>. Therefore approximately 590 subjects will be randomly selected for BICR. All randomized subjects who have {baseline CT/MRI scan and at least one post-baseline CT/MRI scan} OR {baseline bone scan and at least one post-baseline bone scan} will be eligible for the random sample generation.

All scans will be collected and stored in a central location so that a valid audit can be performed using independent centralized review of blinded radiographic scans. Assuming a compelling and clinically meaningful investigator-assessed treatment effect size is present, based on the Independent Data Monitoring Committee (IDMC) review and recommendation, the upper limit of the 2-sided 95% confidence interval for the overall estimated log HR by LE based on the audited subset can be estimated by Equation (3) of Dodd et al. Specifically, the estimated overall log HR by LE is expressed as

$$\widetilde{\theta}_{c} = \hat{\theta}_{CA} + \hat{\rho}\sqrt{\delta}(1-\delta)\sqrt{\frac{\hat{V}_{CA}}{\hat{V}_{L}}}(\hat{\theta}_{L\overline{A}} - \hat{\theta}_{LA})$$

where,  $\delta$  is the proportion of available audit subjects out of the total randomized subjects.  $\theta_{CA}$  is the log HR) based on BICR assessed rPFS related datasets that are audited.  $\hat{\theta}_{LA}$  is the log (HR) based on investigator's assessed rPFS related datasets that are audited.  $\hat{\theta}_{L\overline{A}}$  is log (HR) based on the investigator's assessed rPFS related datasets that are not audited.  $\hat{V}_L$  is the variance estimate of log HR based on the overall investigator's assessed rPFS related datasets. The  $\hat{\rho}$  is correlation coefficient between  $\hat{\theta}_{CA}$  and  $\hat{\theta}_{LA}$  that will be estimated using bootstrap method with 6000 samples.

Let  ${}^{\gamma_c}$  be the upper bound of one-sided (1- $\alpha$ /2) CI for  $\widetilde{\theta_c}$ , and CIF be the clinical irrelevance factor. Based on a minimally relevant improvement in rPFS, it is set that CIF =  $\log(1) = 0$  for a hazard ratio of 1 for the proposed audit plan. If this upper limit of the overall estimated log HR by BICR is below 0 or the overall estimated HR by BICR is below 1, then the concordance of the estimates by LE and BICR will be confirmed. Kaplan-Meier methodology will be used to compare the rPFS curves derived from LE and BICR of the audited subset of patients to demonstrate no evidence of bias.

IDMC will review the audit findings and make recommendations. The audit analysis will be coordinated through the independent SSG statistician for the IDMC review. Therefore, all investigators, study team, and the central reviewer will remain blinded to treatment assignment until the IDMC reviews the audit findings and confirms that no bias is present in the investigator review. If bias is considered present, a complete-case of BICR will be considered.

A sensitivity audit analysis will be performed using PhRMA method (Amit et.al., EJC 2011)<sup>[7]</sup>. The method can be found in Attachment 2.

## **5.2.4.** Other Analyses related to Primary Endpoint

#### **Subgroup Analysis**

To assess the consistency of treatment benefit with respect to the primary efficacy endpoint of rPFS within the important subgroups defined in Section 2.4, a univariate non-stratified proportional hazard model will be fitted to evaluate the treatment effect within each subgroup, the hazard ratio and 95% confidence interval will be estimated. Forest plots will also be provided.

#### **Multivariate Analysis**

To evaluate the treatment effect when controlling for clinically meaningful factors at baseline, multivariate Cox regression analysis, adjusting for important selected prognostic factors, will be performed as supportive analysis, if appropriate. The adjusted hazard ratio and its 95% confidence interval for treatment and each factor will be provided. The following baseline covariates may be considered for inclusion in the model:

- Visceral metastases (IWRS: presence, absence)
- ECOG performance status at randomization (IWRS: 0, 1)
- PSA (continuous)
- Lactate dehydrogenase
- Alkaline phosphatase
- Hemoglobin
- Bone metastasis only (yes, no)
- Age

#### **Clinical Progression**

As an exploratory analysis, Time from rPFS to clinical progression (CP) may be summarized by treatment arm if sufficient number of subjects reaches CP during the study. Clinical Progression is defined in Section 5.4.2:

## **Other Analysis**

The number of patients who remained on study drug beyond radiographic progression and the duration that they remained on study drug may be summarized by treatment arm if sufficient number of subjects belong to this category.

## 5.3. Secondary Endpoints

The analyses of the secondary endpoints will be performed at the time of the first interim analysis of OS.





The above procedure will control the familywise type I error rate at 0.05 [5].



## **5.3.1.** Definition

• Overall survival (OS) is defined as the time from randomization to the date of death from any cause. Subjects who are alive at the time of the analysis will be censored on the last known date that they were alive.

- Time to chronic opioid use (defined as administration of additional opioid analgesics lasting for ≥ 3 weeks for oral; or for ≥ 7 days for non-oral formulation) is defined as the time from randomization to the first date of chronic opioid use. Subjects who did not meet the definition of chronic opioid use at the time of the analysis will be censored on the last known date with no chronic opioid use.
- Time to initiation of cytotoxic chemotherapy is defined as the time from randomization to the date of initiation of cytotoxic chemotherapy. Subjects who did not initiate cytotoxic chemotherapy at the time of the analysis will be censored on the last known alive date.
- Time to pain progression is a composite endpoint, defined as the time from the date of randomization to the first date a subject experiences: A. {an increase by 2 points from baseline in the BPI-SF worst pain intensity score (BPI3) observed at 2 consecutive evaluations ≥ 3 weeks apart}, or B. {initiation of chronic opioids as defined in Time to chronic opioid use above}, whichever occurs first.

Given the fact that BPI-SF will be implemented during the 7-day period leading to each assessment cycle (including Day 1 of the cycle), non-missing daily BPI3 pain scores from the 7-day collection with minimum of 1 day entries is averaged to be evaluated if an increase by 2-point has occurred.

Subjects with no pain progression at the time of analysis will be censored at the last known date of no progression. All sensitivity analyses for this endpoint are included in a separate SAP for PRO analysis.

For all these time-to-events endpoints, subjects with no on-study assessment or no baseline assessment will be censored on the date of randomization. Additionally, sensitivity analyses will be performed for time to chronic opioid use and time to pain progression endpoints, the initiation of anti-cancer subsequent therapy will be used to censor the event after the therapy.

## 5.3.2. Analysis Methods

The testing of these secondary efficacy endpoints will be based on the stratified log rank test. Secondary efficacy endpoints will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. Cox proportional hazard models will be used to estimate the HR and its 95% confidence interval.

#### 5.3.3. Additional Analysis for OS

The following sensitivity analyses for the OS may be carried out as appropriate if it is deemed useful to aid in the interpretation of the results.

#### **Subgroup Analysis**

To assess the consistency of treatment benefit with respect to the primary efficacy endpoint of rPFS within the important subgroups defined in Section 2.4, a univariate non-stratified proportional hazard model will be fitted to evaluate the treatment effect within each subgroup, the hazard ratio and 95% confidence interval will be estimated. Forest plots will also be provided.

Examination of overall survival may be performed to compare patients who received a concurrent androgen receptor inhibitor and abiraterone with patients who received abiraterone followed by enzalutamide after discontinuation of study treatment. This is to evaluate the possibility of reduced efficacy of enzalutamide after abiraterone failure, the issue of whether concomitant abiraterone + 2nd generation antiandrogen is superior to a sequential approach (abiraterone followed by enzalutamide in the U.S.).

## **Multivariate Analysis**

Multivariate analysis of OS adjusting for baseline prognostic factors will be performed similarly as rPFS outlined in Section 5.2.5. The adjusted hazard ratio and its 95% confidence interval for treatment and each factor will be provided. The results may be used to support the findings obtained from the primary analysis.

## **Sensitivity Analysis for OS**

A large number of subjects are expected to receive subsequent anti-cancer therapies after discontinuing study treatment, the following analyses may be used, if appropriate, in estimating the true treatment effect on OS:

- Inverse Probability Censoring Weighted (IPCW) log-rank test as described by Cole and Hernan<sup>[9]</sup>
- Using a time-dependent Cox regression; the HR prior to receiving subsequent anti-cancer therapy and after will be estimated, the associated 95% CI will be calculated.

## 5.4. Other Efficacy Analyses

#### 5.4.1. Definition

Other efficacy endpoints are defined in Table 3.

**Table 3: Other Endpoints** 

| Table 5. Oth | ici Enaponits | |
|---|---|---|
| Endpoint | Description | Analysis Population |
| Time to deterioration of ECOG PS | Primary Analysis: Defined as the time from randomization to the date of deterioration in ECOG PS grade (increase by at least 1 grade from baseline with confirmation at least 4 weeks apart). | ITT Population |
| | Sensitivity Analysis: the deterioration in ECOG PS grade is defined as the following: from 0 or 1 increase to 2 or above; or from 2 increase to 3. | |
| Time to<br>symptomatic<br>skeletal-related<br>event (TTSSRE) | The time from randomization to first occurrence of one of the following: Use of external beam radiation therapy (EBRT) to relieve skeletal symptoms The occurrence of new symptomatic bone fractures (cancerrelated: vertebral or non-vertebral) The occurrence of tumor-related spinal cord compression Need for tumor-related orthopedic surgical intervention | ITT Population |
| | Subjects who have no symptomatic skeletal-related event (SSRE) at the time of analysis will be censored at the last known on-study date of no SSRE. | |
| Objective response rate | Objective response rate defined as the proportion of subjects with measurable disease achieving a complete or partial response according to modified RECIST 1.1. | Subjects with measurable disease at Baseline |

| Table 3: Otl | her Endpoints | |
|---|---|---|
| Endpoint | Description | Analysis Population |
| Duration of response | Duration of response in subjects with measurable disease (based on modified RECIST 1.1) is defined from the time of documented response to the first date of documented progression. Subjects who have not been administered with cytotoxic chemotherapy at the time of analysis will be censored on the last known date of no cytotoxic chemotherapy. | Subjects with CR or PR |
| Health related- | The patient-reported outcomes will include the following: | ITT Population |
| Quality of Life<br>(HRQOL) | <ul> <li>BPI-SF: worst pain intensity score (Item 3), pain interference score (combining Items 9a-9g), and average pain (average of Items 3-6) that are based on average of 7-day diary.</li> <li>FACT-P: FACT-P total score, each subscale score (PWB, SFWB, EWB, FWB, FACT-G, PCS), TOI, PRS, and</li> </ul> | |
| | <ul> <li>FAPSI-8.</li> <li>EQ-5D-5L: 5 domain levels and VAS score; Health Utility Index (HUI).</li> <li>See PRO SAP for the PRO endpoint definition and analysis methods.</li> </ul> | |
| Time to analgesic progression | The time from randomization to the first date of an increase in analgesic usage score of one level increase from baseline observed at 2 consecutive evaluation ≥4 weeks apart. Subjects with no analgesic progression at the time of analysis will be censored on the last known date the subject was known to have not progressed. | ITT Population |
| Time to PSA progression | The time from randomization to the first date of documented PSA progression per PCWG2 criteria. Subjects with no PSA progression at the time of analysis will be censored on the last known date with no progression. | ITT Population |
| PSA response<br>Rate | Proportion of subjects achieving a PSA decline of ≥50% according to PCWG2 criteria. | ITT Population |
| Progression-free<br>survival on first<br>subsequent<br>therapy (PFS2) | PFS2 is defined as time from randomization to the date of first progression (radiographic, clinical, or PSA progression) on the first subsequent therapy or death from any cause, whichever occurs first | ITT population |

| Table 3: | Other 1 | <b>Endpoints</b> |
|----------|---------|------------------|
|----------|---------|------------------|

| Endpoint | Description | Analysis Population |
|---|---|---|
| Time to clinical progression | Description A composite endpoint is defined as time from randomization to first occurrence of one of the following: 1. deterioration in ECOG PS to grade 3; 2. need to initiate any of the following: a. alternative anti-cancer therapy (systemic), b. the use of external beam radiation therapy for tumor related symptoms c. the need for tumor-related surgical intervention/procedure; d. the need for chronic opioid analgesics (per protocol | Analysis Population ITT population |
| | <ul><li>definition);</li><li>e. cancer-related symptomatic events of clear clinical significance.</li></ul> | |
| | If no event was observed, subject will be censored at the last known alive date. | |
| | In addition, a sensitivity analysis excluding the component of deterioration of ECOG performance status from the composite endpoint will be performed. | |

## 5.4.2. Analysis Methods

Analyses of the other endpoints (except for HRQOL measures) will be performed on the ITT population, unless otherwise specified. Time-to-event endpoints and endpoints with binary outcome will be carried out as described above. HRQOL measures related endpoints, and analysis strategies are described in Section 5.4.3 below.

## 5.4.3. Patient Reported Outcome (PRO)

A separate statistical analysis plan will be provided for PRO data.

#### 6. SAFETY

#### 6.1. Adverse Events

Subjects will be assessed for adverse events (AEs) at each monthly clinic visit while on the study. Adverse events will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 and coded to preferred term and system organ class (SOC) using the MedDRA version 20.0.

All AEs reported during the AE reporting period (inclusive of the 30-day post last dose of study drug period) will be considered as treatment-emergent adverse events and will be summarized by treatment group as treated using all subjects in the safety population.

For each treatment group, adverse event incidence rates will be summarized with frequency and percentage by SOC and preferred term, with all subjects treated in that treatment group as the denominator, unless otherwise specified. In addition, AE incidence rates will also be summarized by severity and relationship to study drug. Treatment-related AEs are those judged by the Investigator to be at least possibly related to the blinded study drug. Subjects with multiple occurrences of events will only

be counted once at the maximum severity to study drug for each preferred team, SOC, and overall. Deaths that occur within 30 days after the last dose of study drug are defined as on-study deaths.

Summary tables of the following AEs will be provided:

- Overall summary of AEs: the number and percentage of subjects who experienced any AE, Grade 3/4 AEs, any serious adverse event (SAE), any treatment-related AE, treatment related Grade 3/4 AE, any treatment-related SAE, AE leading to treatment discontinuation, related AE leading to treatment discontinuation, AE leading to death, related AE leading to death, and all deaths within 30 days of last dose
- All AEs by SOC and preferred term (for all AEs and for most frequent AEs (reported in ≥ 5% of subjects))
- All AEs by SOC, preferred term, and toxicity grade
- All AEs by decreasing frequency of preferred term
- Grades 3 or 4 AEs by SOC and preferred term
- Treatment-related AEs by SOC and preferred term
- Treatment-related AEs by SOC, preferred term, and toxicity grade
- Treatment-related Grades 3 or 4 AEs by SOC and preferred term (for all Grades 3 and 4 AEs and for Grades 3 and 4 most frequent AEs (reported ≥ 1% of subjects))
- AEs that led to study drug discontinuation by SOC and preferred term. Study drug discontinuation will be determined from the End of Treatment CRF (where reason for termination is "Adverse Event") and the specific AE will be determined from the AE CRF page (where action taken is "Withdrawn from Study")
- AEs that led to study drug discontinuation by SOC, preferred term, and toxicity grade
- All SAEs by SOC and preferred term
- All SAEs by SOC, preferred term, and toxicity grade
- Deaths will be summarized by time period (on-study vs. during follow-up) and cause of death.

The incidence of AEs of special interest will be summarized by category and preferred term. Adverse Events of Special Interest for apalutamide + AAP include:

- Seizure
- Fall (relationship to syncope or dizziness will be assessed)
- Hypothyroidism
- Skin Rash
- Fracture (relationship to medical history or adverse event of osteoporosis or osteopenia will be assessed along with relationship of AE of change in weight and use of bone targeted agents at doses for treatment of either osteoporosis or metastatic disease that were initiated prior to or following the event)
- Osteoporosis/Osteopenia excluding fracture
- Rhabdomyolysis/Myopathy
- Cardiac disorders (ischaemic heart disease, arrhythmia, cardiac failure, and other cardiac disorders)

- Hepatotoxicity
- Allergic alveolitis
- Hypertension
- Hypokalemia
- Fluid retention/oedema

Note that fall is a single preferred term, all other categories are comprised of a group of preferred terms. A listing of preferred terms that comprise the groupings are provided in Attachment 1.

The AEs of clinical importance will be summarized by category and preferred term. Adverse events of clinical importance include: Diabetes and Cognitive Deficits, which were identified based on previous experience with apalutamide. A listing of the single preferred terms that comprise the groupings are provided in Attachment 1.

Subject listings of all Grades 3 or 4 AEs, all SAEs, AEs that led to study drug discontinuation, and all deaths will be provided as well.

Narratives will be written for the following subjects in the final clinical study report:

- Deaths within 30 days of the last dose of study drug
- Subjects who have serious adverse event
- Subjects who discontinue study drug due to adverse events
- Subjects who experience AEs of special interest of seizure (any grade)
- Other treatment-emergent AEs of special interest (grade 3 or higher) including skin rash, fractures, fall, and hypothyroidism
- Grade 3 or higher major adverse cardiovascular events (MACE) to include ischemic heart disease, cardiac failure, cerebrovascular disease, and arrhythmias.

## **6.2.** Clinical Laboratory Tests

Only data collected by the central laboratory will be summarized. Local laboratory data collected during study for the purposes of planning treatment administration, dose modification, or monitoring adverse events, will not be summarized.

Normal ranges will be used to identify values that are outside the normal ranges and abnormal laboratory results will be graded according to the NCI CTCAE Version 4.03.

A shift summary of baseline grade vs worst post-baseline CTCAE grade will be presented, as appropriate for selected parameters. For each laboratory parameter, the baseline laboratory value will be defined as the last laboratory value collected on or prior to the date of the first dose of study drug.

A listing of subjects who develop toxicities of Grade  $\geq 3$  will be provided for each lab parameter.

Subjects meeting lab criteria for eDISH (Evaluation of Drug Induced Serious Hepatotoxicity) will be listed. eDISH is defined as 1) Elevated ALT or AST at any time. That is, max (ALT/ULN) > 3 or max (AST/ULN) > 3. 2) Elevated TBL at any time. That is, max (TBL/ULN) > = 2.

## 6.3. Vital Signs and Physical Examination Findings

Baseline vital sign (temperature, blood pressure (systolic and diastolic), respiration rate, and heart rate) will be summarized by treatment group. Only blood pressure and body weight are reported during treatment phase. Subjects with markedly abnormalities in blood pressure as compared to baseline will be summarized according to the following categories defined below.

| Parameter | Criteria for Markedly Abnormality |
|---|---|
| Systolic Blood | Absolute result < 90 mmHg and decrease from baseline > 20 mmHg |
| Pressure | Absolute result > 160 mmHg and increase from baseline > 20 mmHg |
| Diastolic Blood | Absolute result < 50 mmHg and decrease from baseline > 10 mmHg |
| Pressure | Absolute result > 100 mmHg and increase from baseline > 10 mmHg |
| | 5 - < 10% weight loss from baseline |
| Weight (kg)a | 10 - < 20% weight loss from baseline |
| | >= 20% weight loss from baseline |

# 6.4. Electrocardiogram

Electrocardiograms (ECGs) (12-lead) will only be recorded at screening, and no QT data are collected. Abnormalities reported at screening will be summarized.

## 7. PHARMACOKINETICS

Pharmacokinetic assessment (trough PK samples) will be per protocol. Pre-dose blood samples (up to 1 hour prior to on-site study drugs administration) will be drawn as described in the Laboratory Manual on Day 1 of Cycles 1, 2, 3, 4, 5 and 6.

Analyses on PK data will be conducted and reported separately.

#### 8. BIOMARKERS

A pre-defined biomarker signature based on the mRNA expression of component genes such as (FLH1, MT1E, SF1 and STARD4) will be evaluated. For each of the subjects with the biomarker sample collected and evaluated, expression status of the biomarker signature (i.e. Positive/Negative) will be assigned. If adequate data is available, efficacy analysis (including but may not be limited to: rPFS, time to PSA progression, overall survival, PSA response rate, and objective response rate) will be performed within the biomarker signature positive and biomarker signature negative subgroups comparing apalutamide plus AAP versus AAP alone.

Other exploratory biomarker analysis may also be performed to assess the association of the rest of the biomarkers with clinical response or time-to-event endpoints using appropriate statistical methods, (such as analysis of variance [ANOVA], categorical or survival models), depending on the endpoints. Analyses may be performed within and between each treatment group. Other clinical covariates (such as baseline tumor characteristics and patient demographics) may also be included in the model. Results of these exploratory analyses will be presented in separate technical reports.

# 9. MEDICAL RESOUURCE UTILIZATION

Medical resource utilization will be descriptively summarized by treatment group. This report will be prepared separately and will not be a part of the clinical study report.

## **REFERENCES**

- 1. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: Revised RECIST guideline (version 1.1). Eur J Cancer 45: 228-47, 2009.
- 2. Scher HI, Halabi S, et al. Design and End Points of Clinical Trials for Patients With Progressive Prostate Cancer and Castrate Levels of Testosterone: Recommendations of the Prostate Cancer Clinical Trials Working Group. Journal of Clinical Oncology, Vol 26, No 7, 1148-1159, 2008.
- 3. Wang SK and Tsiatis AA (1987). Approximately optimal one-parameter boundaries for group sequential trials. Biometrics, 43, 193-199.
- 4. Dmitrienko, A., Tamhane, A., Wiens, B. (2008). General multistage gatekeeping procedures. Biometrical Journal. 50, 667-677.
- 5. Kaplan EL and Meier P. Nonparametric estimation from incomplete observations. J Am Stat Assoc 1958; 53:457-81
- 6. Dodd LE, Korn EL, et al. An audit strategy for progression-free survival. Biometrics 2011; 67, 1092-1099
- 7. Amit O, Mannino F, et al. Blinded independent central review of progression in cancer clinical trials: Results from a meta-analysis. European Journal of Cancer 2011, 47, 1772-1778
- 8. Zhang JJ, Zhang L, Chen H, Murgo AJ, Dodd LE, Pazdur R, and Sridhara R Assessment of Audit Methodologies for Bias Evaluation of Tumor Progression in Oncology Clinical Trials. Clin Cancer Res 2013;19:2637-2645.
- 9. Robins JM and Tsiatis AA. Correcting for non-compliance in randomized trials using Rank Preserving Structural Failure Time models. Commun Statist Theory Meth 1991; 20:2609-2631
- 10. Cole SR and Hernán MA Adjusted survival curves with inverse probability weights. Computer Methods and Programs in Biomedicine 2004; 75:45-49
- 11. Branson M and Whitehead J. Estimating a treatment effect in survival studies in which patients switch treatment. Statistical Medicine 2002; 21, 2449-2463.
- 12. Cella D, Nichol MB, et al. Estimating Clinically Meaningful Changes for the Functional Assessment of Cancer Therapy Prostate: Results from a Clinical Trial of Patients with Metastatic Hormone-Refractory Prostate Cancer. *Value in Health* 12(1): 124-129, 2009
- 13. Cella D, Zarari MJ, et al. Epoetin Alfa Treatment Results in Clinically Significant Improvements in Quality of Life in Anemic Cancer Patients when Referenced to the General Population. *JCO* 21(2): 366-373, 2003

28

#### Attachment 1: Audit Analysis Using Amit's Method

To confirm that the investigator review is not biased in favor of the experimental arm for primary analysis of rPFS, a sensitivity audit analysis will be performed based on the publication of Amit et al <sup>[7]</sup>.

Based on the 590 subjects randomly selected for BICR, the audit will use calculations of early discrepancy rates (EDR) and late discrepancy rates (LDR) for each treatment group to determine whether bias is present in the investigator assessments. For this study, bias will be considered present in the investigator review if the EDR in the experimental arm is lower than EDR in the control arm, or LDR in the experimental arm is higher than LDR in the control arm. Specifically, Table 4 shows the agreement between Blinded Independent Central Review and Investigator Review.

Table 4: Blinded Independent Central Review versus Investigator Review of Disease Progression

| _ | Blinded Independent Central Review | |
|-----------------|------------------------------------|-------|
| | PD | No PD |
| Investigator PD | a = a1 + a2 + a3 | b |
| No PD | С | d |

- a1: number of agreements on timing and occurrence of PD.
- a2: number of times investigator declares PD later than Central Review.
- a3: number of times investigator declares PD earlier than Central Review.

The early discrepancy rate (EDR) of the investigator review is defined as:

$$EDR = \frac{b + a_3}{a + b}$$

The late discrepancy rate (LDR) of the investigator review is defined as:

$$LDR = \frac{c + a_2}{b + c + a_2 + a_3}$$

Note the EDR and LDR represent the frequency with which the investigator review declares progression earlier than independent review (EDR) and the frequency with which the investigator review declares progression later than independent review (LDR).

Bias will be considered present in the investigator review if

EDR (experimental arm) < EDR (control arm) indicating the EDR in the experimental arm is lower than EDR in the control arm,

or

LDR (experimental arm) > LDR (control arm) indicating LDR in the experimental arm is higher than LDR in the control arm.

The final determination of EDR and LDR for each treatment arm and interpretation of the findings will be coordinated by the independent SSG statistician for IDMC. Therefore, all

investigators, Company personnel, and the central reviewer will remain blinded to treatment assignment until the IDMC reviews the audit findings.

## Attachment 2: Adverse Events of Special Interest or Clinical importance

The search criteria of adverse event(s) of interest (AEOI) are based on adverse event preferred terms from MedDRA Version 20.0 dictionary.

Most categories are based on a MedDRA SMQ but if one does not exist a compilation of terms that reflect the event will be proposed for extraction and analysis of the data. Each of these events is defined below:

| Adverse Event of Special Interest Category=Seizure Search Criteria Category= Selected PTs | |
|---|---|
| Acquired epileptic aphasia | Hypoglycaemic seizure |
| Acute encephalitis with refractory, repetitive partial seizures | Hyponatraemic seizure |
| Alcoholic seizure | Idiopathic generalised epilepsy |
| Amygdalohippocampectomy | Lafora's myoclonic epilepsy |
| Aspartate-glutamate-transporter deficiency | Lennox-Gastaut syndrome |
| Atonic seizures | Migraine-triggered seizure |
| Atypical benign partial epilepsy | Molybdenum cofactor deficiency |
| Aura | Myoclonic epilepsy |
| Automatism epileptic | Myoclonic epilepsy and ragged-red fibres |
| Autonomic seizure | Narcolepsy |
| Baltic myoclonic epilepsy | Partial seizures |
| Benign rolandic epilepsy | Partial seizures with secondary generalisation |
| Biotinidase deficiency | Petit mal epilepsy |
| CSWS syndrome | Polymicrogyria |
| Change in seizure presentation | Post stroke epilepsy |
| Clonic convulsion | Post stroke seizure |
| Complex partial seizures | Post-traumatic epilepsy |
| Convulsion prophylaxis | Postictal headache |
| Convulsions local | Postictal paralysis |
| Convulsive threshold lowered | Postictal psychosis |
| Corpus callosotomy | Postictal state |
| Deja vu | Preictal state |
| Double cortex syndrome | Psychomotor seizures |
| Dreamy state | Schizencephaly |
| Drop attacks | Seizure |
| Drug withdrawal convulsions | Seizure anoxic |

| Epilepsy | Seizure cluster |
|---|---|
| Epileptic aura | Seizure like phenomena |
| Epileptic psychosis | Severe myoclonic epilepsy of infancy |
| Febrile convulsion | Simple partial seizures |
| Febrile infection-related epilepsy syndrome | Status epilepticus |
| Foaming at mouth | Sudden unexplained death in epilepsy |
| Focal dyscognitive seizures | Temporal lobe epilepsy |
| Frontal lobe epilepsy | Tongue biting |
| Generalised non-convulsive epilepsy | Tonic clonic movements |
| Generalised tonic-clonic seizure | Tonic convulsion |
| Glucose transporter type 1 deficiency syndrome | Tonic posturing |
| Hemimegalencephaly | Topectomy |
| Hyperglycaemic seizure | Uncinate fits |

| Search Criteria Category= Selected PTs | |
|--------------------------------------------|-----------------------------|
| Acquired epidermolysis bullosa | Noninfective conjunctivitis |
| Acute generalised exanthematous pustulosis | Oculomucocutaneous syndrome |
| Administration site hypersensitivity | Oral mucosal blistering |
| Administration site rash | Oral mucosal exfoliation |
| Administration site recall reaction | Oral papule |
| Administration site urticaria | Oropharyngeal blistering |
| Application site rash | Papule |
| Blau syndrome | Paraneoplastic rash |
| Blister | Pemphigoid |
| Blister rupture | Pemphigus |
| Bullous impetigo | Penile exfoliation |
| Butterfly rash | Perineal rash |
| Catheter site rash | Pogosta disease |
| Conjunctivitis | Rash |
| Corneal exfoliation | Rash erythematous |
| Cutaneous vasculitis | Rash follicular |
| Dermatitis bullous | Rash generalised |
| Dermatitis exfoliative | Rash macular |
| Dermatitis exfoliative generalised | Rash maculo-papular |
| Drug eruption | Rash maculovesicular |

Rash morbilliform

Drug reaction with eosinophilia and systemic symptoms

| Epidermal necrosis | Rash papular |
|---|---|
| Epidermolysis | Rash papulosquamous |
| Epidermolysis bullosa | Rash pruritic |
| Eruptive pseudoangiomatosis | Rash pustular |
| Erythema multiforme | Rash rubelliform |
| Exfoliative rash | Rash scarlatiniform |
| Eyelid rash | Rash vesicular |
| Familial cold autoinflammatory syndrome | Sea bather's eruption |
| Fixed drug eruption | Skin erosion |
| Genital rash | Skin exfoliation |
| Genital ulceration | Skin necrosis |
| HLA-B*1502 assay positive | Skin reaction |
| HLA-B*5801 assay positive | Skin swelling |
| Hyper IgD syndrome | Staphylococcal scalded skin syndrome |
| Hypopharyngeal synechiae | Stevens-Johnson syndrome |
| Implant site rash | Stoma site rash |
| Incision site rash | Stomatitis |
| Infusion site rash | Symmetrical drug-related intertriginous and flexural exanthema |
| Injection site rash | Systemic lupus erythematosus rash |
| Instillation site rash | Tongue exfoliation |
| Lip exfoliation | Toxic epidermal necrolysis |
| Lupus miliaris disseminatus faciei | Toxic skin eruption |
| Medical device site rash | Urticaria |
| Mouth ulceration | Urticaria papular |
| Mucocutaneous rash | Vaccination site rash |
| Mucocutaneous ulceration | Vaginal exfoliation |
| Mucosa vesicle | Vaginal ulceration |
| Mucosal erosion | Vascular access site rash |
| Mucosal exfoliation | Vessel puncture site rash |
| Mucosal necrosis | Viral rash |
| Mucosal ulceration | Vulval ulceration |
| Nikolsky's sign | Vulvovaginal rash |
| Nodular rash | Vulvovaginal ulceration |
| Adverse Event of Special Interest Category=Hypothyroidism Search Criteria Category= Selected PTs (SMQ) | |
| Anti-thyroid antibody | Secondary hypothyroidism |
|---|---|
| Anti-thyroid antibody positive | Silent thyroiditis |
| Atrophic thyroiditis | Tertiary hypothyroidism |
| Autoimmune hypothyroidism | Thyroglobulin absent |
| Autoimmune thyroid disorder | Thyroglobulin decreased |
| Autoimmune thyroiditis | Thyroid atrophy |
| Blood thyroid stimulating hormone increased | Thyroid hemiagenesis |
| Butanol-extractable iodine decreased | Thyroid hormone replacement therapy |
| Congenital hypothyroidism | Thyroid therapy |
| Congenital thyroid disorder | Thyroidectomy |
| Free thyroxine index decreased | Thyroiditis |
| Generalised resistance to thyroid hormone | Thyroiditis acute |
| Hashimoto's encephalopathy | Thyroiditis chronic |
| Hypothyroidic goitre | Thyroiditis fibrous chronic |
| Hypothyroidism | Thyroiditis subacute |
| Iodine uptake decreased | Thyroxin binding globulin increased |
| Myxoedema | Thyroxine decreased |
| Myxoedema coma | Thyroxine free decreased |
| Polyglandular autoimmune syndrome type II | Thyroxine therapy |
| Polyglandular autoimmune syndrome type III | Transient hypothyroxinaemia of prematurity |
| Post procedural hypothyroidism | Tri-iodothyronine decreased |
| Primary hypothyroidism | Tri-iodothyronine free decreased |
| Protein bound iodine decreased | Tri-iodothyronine uptake increased |
| Reverse tri-iodothyronine decreased | |
| Adverse Event of Special Interest Category=Fall | |
| Search Criteria Category= Selected PTs | |
| Fall | |
| Adverse Event of Special Interest=Fracture | |
| Search Criteria Category= Selected PTs | |
| Acetabulum fracture | Hand fracture |
| Ankle fracture | Hip fracture |
| Atypical femur fracture | Humerus fracture |
| Atypical fracture | Ilium fracture |
| Avulsion fracture | Impacted fracture |
| Cervical vertebral fracture | Internal fixation of fracture |

| Chance fracture | Jaw fracture |
|---|---|
| Clavicle fracture | Limb fracture |
| Closed fracture manipulation | Loss of anatomical alignment after fracture reduction |
| Comminuted fracture | Lower limb fracture |
| Complicated fracture | Lumbar vertebral fracture |
| Compression fracture | Multiple fractures |
| Costal cartilage fracture | Open fracture |
| Craniofacial fracture | Open reduction of fracture |
| Elevation skull fracture | Open reduction of spinal fracture |
| Epiphyseal fracture | Osteochondral fracture |
| External fixation of fracture | Osteoporotic fracture |
| Facial bones fracture | Patella fracture |
| Femoral neck fracture | Pelvic fracture |
| Femur fracture | Periprosthetic fracture |
| Fibula fracture | Pubis fracture |
| Foot fracture | Radius fracture |
| Forearm fracture | Rib fracture |
| Fracture | Sacroiliac fracture |
| Fracture debridement | Scapula fracture |
| Fracture delayed union | Skull fracture |
| Fracture displacement | Skull fractured base |
| Fracture malunion | Spinal compression fracture |
| Fracture nonunion | Spinal fracture |
| Fracture of clavicle due to birth trauma | Spinal fusion fracture |
| Fracture of penis | Sternal fracture |
| Fracture pain | Stress fracture |
| Fracture reduction | Surgical fixation of rib fracture |
| Fracture treatment | Thoracic vertebral fracture |
| Fractured coccyx | Tibia fracture |
| Fractured ischium | Torus fracture |
| Fractured maxilla elevation | Traumatic fracture |
| Fractured sacrum | Ulna fracture |
| Fractured skull depressed | Upper limb fracture |
| Fractured zygomatic arch elevation | Wrist fracture |
| Greenstick fracture | |

Adverse Event of Special Interest Category=Ischaemic Heart Disease

| Search Criteria Category= Selected PTs | |
|---|---|
| Acute coronary syndrome | Electrocardiogram ST segment depression |
| Acute myocardial infarction | Electrocardiogram ST segment elevation |
| Angina pectoris | Electrocardiogram ST-T segment abnormal |
| Angina unstable | Electrocardiogram ST-T segment depression |
| Anginal equivalent | Electrocardiogram ST-T segment elevation |
| Arteriogram coronary abnormal | Electrocardiogram T wave abnormal |
| Arteriosclerosis coronary artery | Electrocardiogram T wave inversion |
| Arteriospasm coronary | Exercise electrocardiogram abnormal |
| Blood creatine phosphokinase MB abnormal | Exercise test abnormal |
| Blood creatine phosphokinase MB increased | External counterpulsation |
| Blood creatine phosphokinase abnormal | Haemorrhage coronary artery |
| Blood creatine phosphokinase increased | Infarction |
| Cardiac stress test abnormal | Ischaemic cardiomyopathy |
| Cardiopulmonary exercise test abnormal | Kounis syndrome |
| Computerised tomogram coronary artery abnormal | Microvascular coronary artery disease |
| Coronary angioplasty | Myocardial hypoxia |
| Coronary arterial stent insertion | Myocardial infarction |
| Coronary artery bypass | Myocardial ischaemia |
| Coronary artery disease | Myocardial necrosis |
| Coronary artery dissection | Myocardial necrosis marker increased |
| Coronary artery embolism | Myocardial reperfusion injury |
| Coronary artery insufficiency | Myocardial stunning |
| Coronary artery occlusion | Papillary muscle infarction |
| Coronary artery reocclusion | Percutaneous coronary intervention |
| Coronary artery restenosis | Periprocedural myocardial infarction |
| Coronary artery stenosis | Post procedural myocardial infarction |
| Coronary artery thrombosis | Postinfarction angina |
| Coronary bypass thrombosis | Prinzmetal angina |
| Coronary endarterectomy | Scan myocardial perfusion abnormal |
| Coronary no-reflow phenomenon | Silent myocardial infarction |
| Coronary ostial stenosis | Stress cardiomyopathy |
| Coronary revascularisation | Stress echocardiogram abnormal |
| Coronary vascular graft occlusion | Subclavian coronary steal syndrome |
| Dissecting coronary artery aneurysm | Subendocardial ischaemia |
| ECG electrically inactive area | Troponin I increased |
| ECG signs of myocardial infarction | Troponin T increased |

| ECG signs of myocardial ischaemia | Troponin increased |
|---|---|
| Electrocardiogram Q wave abnormal | Vascular graft occlusion |
| Electrocardiogram ST segment abnormal | |
| Adverse Event of Special Interest Category=Cardiac Failure | |
| Search Criteria Category= Selected PTs | |
| Acute left ventricular failure | Dyspnoea paroxysmal nocturnal |
| Acute pulmonary oedema | Ejection fraction decreased |
| Acute right ventricular failure | Heart transplant |
| Artificial heart implant | Hepatic vein dilatation |
| Atrial natriuretic peptide abnormal | Hepatojugular reflux |
| Atrial natriuretic peptide increased | Jugular vein distension |
| Brain natriuretic peptide abnormal | Left ventricular dysfunction |
| Brain natriuretic peptide increased | Left ventricular failure |
| Cardiac asthma | Low cardiac output syndrome |
| Cardiac cirrhosis | Lower respiratory tract congestion |
| Cardiac failure | Myocardial depression |
| Cardiac failure acute | N-terminal prohormone brain natriuretic peptide abnormal |
| Cardiac failure chronic | N-terminal prohormone brain natriuretic peptide increased |
| Cardiac failure congestive | Neonatal cardiac failure |
| Cardiac failure high output | Nocturnal dyspnoea |
| Cardiac index decreased | Obstructive shock |
| Cardiac output decreased | Oedema due to cardiac disease |
| Cardiac resynchronisation therapy | Orthopnoea |
| Cardiac ventriculogram abnormal | Pulmonary congestion |
| Cardiac ventriculogram left abnormal | Pulmonary oedema |
| Cardiac ventriculogram right abnormal | Pulmonary oedema neonatal |
| Cardio-respiratory distress | Radiation associated cardiac failure |
| Cardiogenic shock | Right ventricular dysfunction |
| Cardiomegaly | Right ventricular failure |
| Cardiopulmonary failure | Stroke volume decreased |
| Cardiorenal syndrome | Systolic dysfunction |
| Cardiothoracic ratio increased | Venous pressure increased |
| Central venous pressure increased | Venous pressure jugular abnormal |
| Chronic left ventricular failure | Venous pressure jugular increased |
| Chronic right ventricular failure | Ventricular assist device insertion |

| Statistical Analysis Plan 56021927PCR3001 – Amendment | |
|---|---|
| Cor pulmonale | Ventricular dysfunction |
| Cor pulmonale acute | Ventricular dyssynchrony |
| Cor pulmonale chronic | Ventricular failure |
| Diastolic dysfunction | Wall motion score index abnormal |
| Dilatation ventricular | |
| Adverse Event of Special Interest Category= | =Arrhythmia |
| Search Criteria Category= Selected PTs | |
| Accelerated idioventricular rhythm | Palpitations |
| Arrhythmia supraventricular | Parasystole |

## Arrhythmia supraventricular Parasystole Atrial fibrillation Rebound tachycardia Atrial flutter Respiratory sinus arrhythmia magnitude abnormal Atrial flutter with 1:1 atrioventricular conduction Respiratory sinus arrhythmia magnitude decreased Respiratory sinus arrhythmia magnitude increased Atrial parasystole Atrial tachycardia Retrograde p-waves Bradycardia Rhythm idioventricular Cardiac arrest Sinus tachycardia Cardiac death Sudden cardiac death Cardiac fibrillation Sudden death Cardiac telemetry abnormal Supraventricular extrasystoles Cardio-respiratory arrest Supraventricular tachyarrhythmia Chronotropic incompetence Supraventricular tachycardia ECG P wave inverted Syncope Electrocardiogram P wave abnormal Tachycardia Electrocardiogram RR interval prolonged Tachycardia paroxysmal Electrocardiogram U-wave abnormality Torsade de pointes Electrocardiogram abnormal Ventricular arrhythmia Electrocardiogram ambulatory abnormal Ventricular extrasystoles Ventricular fibrillation Electrocardiogram change Electrocardiogram repolarisation abnormality Ventricular flutter Heart rate abnormal Ventricular parasystole Heart rate decreased Ventricular pre-excitation

Ventricular tachyarrhythmia

Ventricular tachycardia

## **Clinical Importance Category=Diabetes**

Heart rate increased

Loss of consciousness

Junctional ectopic tachycardia

| Search Criteria Category= Selected PTs | |
|---|---|
| ACQUIRED LIPOATROPHIC DIABETES | GLYCOSYLATED HAEMOGLOBIN INCREASED |
| BLOOD 1,5-ANHYDROGLUCITOL DECREASED | HYPERGLYCAEMIA |
| BLOOD GLUCOSE INCREASED | HYPERGLYCAEMIC HYPEROSMOLAR<br>NONKETOTIC SYNDROME |
| DIABETES COMPLICATING PREGNANCY | HYPERGLYCAEMIC SEIZURE |
| DIABETES MELLITUS | HYPERGLYCAEMIC UNCONSCIOUSNESS |
| DIABETES MELLITUS INADEQUATE CONTROL | HYPEROSMOLAR HYPERGLYCAEMIC STATE |
| DIABETES WITH HYPEROSMOLARITY | IMPAIRED FASTING GLUCOSE |
| DIABETIC ARTERITIS | INSULIN RESISTANCE |
| DIABETIC COMA | INSULIN RESISTANCE SYNDROME |
| DIABETIC HEPATOPATHY | INSULIN RESISTANT DIABETES |
| DIABETIC HYPERGLYCAEMIC COMA | INSULIN-REQUIRING TYPE 2 DIABETES MELLITUS |
| DIABETIC HYPEROSMOLAR COMA | KETOACIDOSIS |
| DIABETIC KETOACIDOSIS | KETONURIA |
| DIABETIC KETOACIDOTIC HYPERGLYCAEMIC COMA | KETOSIS |
| DIABETIC METABOLIC DECOMPENSATION | LATENT AUTOIMMUNE DIABETES IN ADULTS |
| FRUCTOSAMINE INCREASED | METABOLIC SYNDROME |
| FULMINANT TYPE 1 DIABETES MELLITUS | MONOGENIC DIABETES |
| GESTATIONAL DIABETES | NEONATAL DIABETES MELLITUS |
| GLUCOSE TOLERANCE IMPAIRED | PANCREATOGENOUS DIABETES |
| GLUCOSE TOLERANCE IMPAIRED IN PREGNANCY | TYPE 1 DIABETES MELLITUS |
| GLUCOSE URINE PRESENT | TYPE 2 DIABETES MELLITUS |
| GLYCOSURIA | TYPE 3 DIABETES MELLITUS |
| GLYCOSURIA DURING PREGNANCY | URINE KETONE BODY PRESENT |
| Clinical Importance Category=Cognitive Deficits | |
| Search Criteria Category= Selected PTs | |
| Amnesia | Disturbance in attention |
| Cognitive disorder | Memory impairment |
| Adverse Event of Special Interest/Clinical Importance Category=Other Cardiac Disorders | |
| Search Criteria Category= Selected PTs | |
| Atrioventricular block | Electrocardiogram QT prolonged |
| Atrioventricular block first degree | Hypertrophic cardiomyopathy |

| | - |
|---|---|
| Bundle branch block left | Left ventricular hypertrophy |
| Cardiac disorder | Long QT syndrome |
| Cardiomyopathy | Metabolic cardiomyopathy |
| Cardiomyopathy acute | Mitral valve disease |
| Cardiomyopathy alcoholic | Non-obstructive cardiomyopathy |
| Chest pain | Restrictive cardiomyopathy |
| Conduction disorder | Sinus arrhythmia |
| Congestive cardiomyopathy | Sinus bradycardia |
| Cytotoxic cardiomyopathy | Sinus node dysfunction |
| Diabetic cardiomyopathy | Viral cardiomyopathy |
| Electrocardiogram QT interval abnormal | Wandering pacemaker |
| Adverse Event of Special Interest Category=Osteoporosis/Osteopenia excluding Fracture | |
| Search Criteria Category= Selected PTs | |
| BONE METABOLISM BIOCHEMICAL MARKER INCREASED | Kyphosis |
| Body height abnormal | N-telopeptide urine increased |
| Body height below normal | Osteocalcin increased |
| Body height decreased | Osteopenia |
| Bone density abnormal | Osteoporosis |
| Bone density decreased | Osteoporosis postmenopausal |
| Bone formation decreased | Osteoporosis prophylaxis |
| Bone formation test abnormal | Post-traumatic osteoporosis |
| Bone loss | Pyridinoline urine increased |
| Bone metabolism disorder | Resorption bone increased |
| Bone resorption test abnormal | Senile osteoporosis |
| C-telopeptide increased | Spinal deformity |
| Deoxypyridinoline urine increased | TARTRATE-RESISTANT ACID PHOSPHATASE DECREASED |
| Hip arthroplasty | Vertebral body replacement |
| Hip surgery | Vertebroplasty |
| Kyphoscoliosis | Wrist surgery |
| Adverse Event of Special Interest Category=Rhabdomyolysis or Myopathy | |
| Search Criteria Category= Selected PTs | |
| Muscle necrosis | Myoglobinuria |
| Myoglobin blood increased | Myopathy |

| Myoglobin blood present | Myopathy toxic |
|---|---|
| Myoglobin urine present | NECROTISING MYOSITIS |
| Myoglobinaemia | Rhabdomyolysis |
| Adverse Event of Special Interest Category=Hypertension | |
| Search Criteria Category= Selected PTs | |
| Accelerated hypertension | Hypertensive cardiomegaly |
| Aldosterone urine abnormal | Hypertensive cardiomyopathy |
| Aldosterone urine increased | Hypertensive crisis |
| Angiotensin I increased | Hypertensive emergency |
| Angiotensin II increased | Hypertensive encephalopathy |
| Angiotensin converting enzyme increased | Hypertensive heart disease |
| Blood aldosterone abnormal | Hypertensive nephropathy |
| Blood aldosterone increased | Labile blood pressure |
| Blood catecholamines abnormal | Labile hypertension |
| Blood catecholamines increased | Malignant hypertension |
| Blood pressure abnormal | Malignant hypertensive heart disease |
| Blood pressure ambulatory abnormal | Malignant renal hypertension |
| Blood pressure ambulatory increased | Maternal hypertension affecting foetus |
| Blood pressure diastolic abnormal | Mean arterial pressure increased |
| Blood pressure diastolic increased | Metabolic syndrome |
| Blood pressure fluctuation | Metanephrine urine abnormal |
| Blood pressure inadequately controlled | Metanephrine urine increased |
| Blood pressure increased | Neurogenic hypertension |
| Blood pressure management | Non-dipping |
| Blood pressure orthostatic abnormal | Norepinephrine abnormal |
| Blood pressure orthostatic increased | Norepinephrine increased |
| Blood pressure systolic abnormal | Normetanephrine urine increased |
| Blood pressure systolic increased | Orthostatic hypertension |
| Catecholamines urine abnormal | PAGE KIDNEY |
| Catecholamines urine increased | Pre-eclampsia |
| Diastolic hypertension | Prehypertension |
| Diuretic therapy | Procedural hypertension |
| Eclampsia | Pseudoaldosteronism |
| Ectopic aldosterone secretion | Renal hypertension |
| Ectopic renin secretion | Renal sympathetic nerve ablation |
| Endocrine hypertension | Renin abnormal |

| Epinephrine abnormal | Renin increased |
|--------------------------------------|-------------------------------------|
| Epinephrine increased | Renin-angiotensin system inhibition |
| Essential hypertension | Renovascular hypertension |
| Gestational hypertension | Retinopathy hypertensive |
| HELLP syndrome | SUPINE HYPERTENSION |
| HYPERTENSIVE CEREBROVASCULAR DISEASE | Secondary aldosteronism |
| HYPERTENSIVE END-ORGAN DAMAGE | Secondary hypertension |
| Hyperaldosteronism | Systolic hypertension |
| Hypertension | Tyramine reaction |
| Hypertension neonatal | Withdrawal hypertension |
| Hypertensive angiopathy | |

## Adverse Event of Special Interest Category=Fluid Retention or Oedema

| Search Criteria Category= Selected PTs | |
|----------------------------------------|------------------------------------|
| Administration site joint effusion | Injection site swelling |
| Administration site oedema | Instillation site oedema |
| Administration site swelling | Joint effusion |
| Amyloid related imaging abnormalities | Joint swelling |
| Application site joint effusion | Lipoedema |
| Application site joint swelling | Local swelling |
| Application site oedema | Localised oedema |
| Application site swelling | Lymphoedema |
| Ascites | Medical device site joint effusion |
| Bone marrow oedema | Medical device site joint swelling |
| Bone marrow oedema syndrome | Mouth swelling |
| Bone swelling | Muscle oedema |
| Brain oedema | Muscle swelling |
| Bronchial oedema | Myocardial oedema |
| COMPRESSION GARMENT APPLICATION | Non-cardiogenic pulmonary oedema |
| Capillary leak syndrome | OROPHARYNGEAL OEDEMA |
| Catheter site oedema | Oedema |
| Cerebral oedema management | Oedema due to renal disease |
| Cervix oedema | Oedema mucosal |
| Compression stockings application | Oedema neonatal |
| Cytotoxic oedema | Oedema peripheral |
| Effusion | Oedematous kidney |

Oesophageal oedema

Elephantiasis nostras verrucosa

| Extensive swelling of vaccinated limb | PERINEPHRIC COLLECTION |
|---|---|
| Fluid overload | PERINEPHRIC OEDEMA |
| Fluid retention | Pelvic fluid collection |
| Gallbladder oedema | Pericardial effusion |
| Gastrointestinal oedema | Peripheral oedema neonatal |
| Generalised oedema | Peripheral swelling |
| Gestational oedema | Pleural effusion |
| Gravitational oedema | Prevertebral soft tissue swelling of cervical space |
| Heat oedema | Puncture site oedema |
| Hydraemia | Reexpansion pulmonary oedema |
| Hydrothorax | Retroperitoneal effusion |
| Hypervolaemia | Retroperitoneal oedema |
| Hypoosmolar state | Scleroedema |
| Implant site oedema | Skin oedema |
| Implant site swelling | Skin swelling |
| Incision site oedema | Spinal cord oedema |
| Incision site swelling | Subdural effusion |
| Infusion site joint effusion | Swelling |
| Infusion site joint swelling | Testicular swelling |
| Infusion site oedema | Vaccination site joint effusion |
| Infusion site swelling | Vaccination site joint swelling |
| Injection site joint swelling | Vasogenic cerebral oedema |
| Injection site oedema | Visceral oedema |
| | Adverse Event of Special Interest Category=Hepatotoxicity |
| Search Criteria Category= Selected PTs | TT COL |
| 5'nucleotidase increased | Hepatitis acute |
| ACUTE ON CHRONIC LIVER FAILURE | Hepatitis cholestatic |
| Abnormal faeces | Hepatitis chronic active |
| Acute graft versus host disease in liver | Hepatitis chronic persistent |
| Acute hepatic failure | Hepatitis fulminant |
| Acute yellow liver atrophy | Hepatitis toxic |
| Alanine aminotransferase abnormal | Hepatobiliary disease |
| Alanine aminotransferase increased | Hepatobiliary scan abnormal |
| Allergic hepatitis | Hepatocellular foamy cell syndrome |
| Ammonia abnormal | Hepatocellular injury |
| | let |

Hepatomegaly

Ammonia increased

| Anorectal varices | Hepatopulmonary syndrome |
|---|---|
| Anorectal varices haemorrhage | Hepatorenal failure |
| Aspartate aminotransferase abnormal | Hepatorenal syndrome |
| Aspartate aminotransferase increased | Hepatosplenomegaly |
| Asterixis | Hepatotoxicity |
| Autoimmune hepatitis | Hyperammonaemia |
| BILIARY DYSPEPSIA | Hyperbilirubinaemia |
| BILIRUBIN EXCRETION DISORDER | Hypercholia |
| BILIRUBIN URINE PRESENT | Hypertransaminasaemia |
| BILIRUBIN URINE PRESENT | Hypoalbuminaemia |
| BIOPSY GALLBLADDER ABNORMAL | INTESTINAL VARICES HAEMORRHAGE |
| Bacterascites | Icterus index increased |
| Bile culture positive | Intestinal varices |
| Bile duct pressure increased | Intrahepatic portal hepatic venous fistula |
| Bile output abnormal | Ischaemic hepatitis |
| Bile output decreased | Jaundice |
| Bile output increased | Jaundice cholestatic |
| Biliary ascites | Jaundice extrahepatic obstructive |
| Biliary cirrhosis | Jaundice hepatocellular |
| Biliary cirrhosis primary | Kayser-Fleischer ring |
| Biliary fibrosis | LIVER DIALYSIS |
| Bilirubin conjugated abnormal | LIVER FUNCTION TEST DECREASED |
| Bilirubin conjugated increased | LIVER FUNCTION TEST INCREASED |
| Bilirubin excretion disorder | Leucine aminopeptidase increased |
| Bilirubinuria | Limy bile syndrome |
| Biopsy bile duct abnormal | Liver and small intestine transplant |
| Biopsy liver abnormal | Liver disorder |
| Blood alkaline phosphatase abnormal | Liver function test abnormal |
| Blood alkaline phosphatase increased | Liver induration |
| Blood bilirubin abnormal | Liver injury |
| Blood bilirubin increased | Liver iron concentration abnormal |
| Blood bilirubin unconjugated increased | Liver iron concentration increased |
| Blood cholinesterase abnormal | Liver operation |
| Blood cholinesterase decreased | Liver palpable |
| Bromosulphthalein test abnormal | Liver sarcoidosis |
| CHILD-PUGH-TURCOTTE SCORE ABNORMAL | Liver scan abnormal |

| Child-Pugh-Turcotte score increased | Liver transplant |
|---|---|
| Cholaemia | Lupoid hepatic cirrhosis |
| Cholangiogram abnormal | Lupus hepatitis |
| Cholecystogram intravenous abnormal | MODEL FOR END STAGE LIVER DISEASE SCORE ABNORMAL |
| Cholecystogram oral abnormal | MODEL FOR END STAGE LIVER DISEASE SCORE INCREASED |
| Cholestasis | Minimal hepatic encephalopathy |
| Cholestatic liver injury | Mitochondrial aspartate aminotransferase increased |
| Cholestatic pruritus | Mixed liver injury |
| Chronic graft versus host disease in liver | Molar ratio of total branched-chain amino acid to tyrosine |
| Chronic hepatic failure | NON-ALCOHOLIC FATTY LIVER |
| Chronic hepatitis | NON-CIRRHOTIC PORTAL HYPERTENSION |
| Coma hepatic | Nodular regenerative hyperplasia |
| Computerised tomogram liver | Non-alcoholic steatohepatitis |
| Cryptogenic cirrhosis | Ocular icterus |
| Deficiency of bile secretion | Oedema due to hepatic disease |
| Diabetic hepatopathy | Oesophageal varices haemorrhage |
| Drug-induced liver injury | PORTAL HYPERTENSIVE COLOPATHY |
| Duodenal varices | PORTAL SHUNT PROCEDURE |
| Endoscopic retrograde cholangiopancreatography abnormal | Parenteral nutrition associated liver disease |
| Endoscopy biliary tract abnormal | Perihepatic discomfort |
| Faeces pale | Peripancreatic varices |
| Foetor hepaticus | Periportal oedema |
| Galactose elimination capacity test abnormal | Peritoneal fluid protein abnormal |
| Galactose elimination capacity test decreased | Peritoneal fluid protein decreased |
| Gallbladder palpable | Peritoneal fluid protein increased |
| Gallbladder varices | Peritoneovenous shunt |
| Gamma-glutamyltransferase abnormal | Pneumobilia |
| Gamma-glutamyltransferase increased | Portal fibrosis |
| Gastric variceal injection | Portal hypertension |
| Gastric variceal ligation | Portal hypertensive enteropathy |
| Gastric varices | Portal hypertensive gastropathy |
| Gastric varices haemorrhage | Portal shunt |
| Glutamate dehydrogenase increased | Portal tract inflammation |
| Graft versus host disease in liver | Portal vein cavernous transformation |
| Granulomatous liver disease | Portal vein dilatation |

| Guanase increased | Portal vein flow decreased |
|---|---|
| HEPATIC STEATO-FIBROSIS | Portal vein pressure increased |
| Haemorrhagic ascites | Portopulmonary hypertension |
| Hepaplastin abnormal | Radiation hepatitis |
| Hepaplastin decreased | Renal and liver transplant |
| Hepatectomy | Retinol binding protein decreased |
| Hepatic artery flow decreased | Retrograde portal vein flow |
| Hepatic atrophy | Reye's syndrome |
| Hepatic calcification | Reynold's syndrome |
| Hepatic cirrhosis | SPLENORENAL SHUNT |
| Hepatic congestion | SPLENORENAL SHUNT PROCEDURE |
| Hepatic encephalopathy | Small-for-size liver syndrome |
| Hepatic encephalopathy prophylaxis | Spider naevus |
| Hepatic enzyme abnormal | Splenic varices |
| Hepatic enzyme decreased | Splenic varices haemorrhage |
| Hepatic enzyme increased | Spontaneous intrahepatic portosystemic venous shunt |
| Hepatic failure | Steatohepatitis |
| Hepatic fibrosis | Stomal varices |
| Hepatic fibrosis marker abnormal | Subacute hepatic failure |
| Hepatic fibrosis marker increased | Total bile acids increased |
| Hepatic function abnormal | Transaminases abnormal |
| Hepatic hydrothorax | Transaminases increased |
| Hepatic hypertrophy | Ultrasound biliary tract abnormal |
| Hepatic infiltration eosinophilic | Ultrasound liver abnormal |
| Hepatic lesion | Urine bilirubin increased |
| Hepatic mass | Urobilinogen urine decreased |
| Hepatic necrosis | Urobilinogen urine increased |
| Hepatic pain | Varices oesophageal |
| Hepatic sequestration | Varicose veins of abdominal wall |
| Hepatic steatosis | WHITE NIPPLE SIGN |
| Hepatic vascular resistance increased | X-ray hepatobiliary abnormal |
| Hepatitis | Yellow skin |
| Adverse Event of Special Interest Category=Hypokalemia | |
| Search Criteria Category= Selected PTs | |
| Blood potassium | Blood potassium decreased |
| Blood potassium abnormal | Hypokalaemia |

| Adverse Event of Special Interest Category=Allergic alveolitis |
|----------------------------------------------------------------|
| Search Criteria Category= Selected PTs |
| Allergic alveolitis |